CLINICAL TRIAL: NCT00701441
Title: The Role of Oxidative Stress in the Cardiovascular Consequences of Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Rami Khayat (Other)
Responsible Party: Sponsor-Investigator, Rami Khayat, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2005H0221
Record Dates: First submitted 2008-05-15; First posted 2008-06-19 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Sleep Apnea
Keywords: sleep apnea,; oxidative stress
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: healthy individuals without OSA: healthy individuals without OSA who are matched in weight and age to the participating OSA patients
- OSA group: Patients in the OSA group receive CPAP for 12 weeks as part of their care. patients with OSA provide measures at baseline and after 12 weeks of CPAP treatment.

SUMMARY:
Obstructive Sleep Apnea (OSA) is the most common sleep disorder affecting up to 9-24 percent of middle aged adults, and is becoming increasingly implicated in the pathogenesis of hypertension, and other cardiovascular disorders. Up to half of patients with OSA have hypertension, and their risk of developing hypertension increases with the increasing severity of Sleep Apnea. Patients with OSA and no hypertension have endothelial dysfunction, which is believed to be the precursor for most cardiovascular disorders.

The upper airway collapse and obstruction that occur in OSA result in a pattern of intermittent hypoxia, that has been shown to be the cause of the hypertension, and endothelial dysfunction found in patients with OSA. Intermittent hypoxia results in oxidative stress, which in turn is linked to the pathogenesis of hypertension and endothelial dysfunction.

This protocol evaluates the role of the oxidative stress in endothelial function and blood pressure in patients with OSA. This is a pilot clinical study that will compare oxidative stress parameters, and endothelial function in patients with OSA before starting treatment with continuous positive airway pressure (CPAP) and 12 weeks post being on CPAP. These patients will be compared to control patients with no history of OSA. the study does not involve assignement to different treatments. All patients will receive the indicated treatment for OSA and measurements will be collected before and 12 weeks after adequate treatment.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is increasingly recognized as a cardiovascular risk factor. OSA is a cause of hypertension and has strong association with atherosclerosis, coronary heart disease, diabetes stroke , and fatal cardiovascular events. Endothelial dysfunction is a preclinical vascular abnormality that predicts subsequent development of vascular disease . Patients with OSA demonstrate endothelial dysfunction in the absence of any manifested vascular disease . The mechanism of endothelial dysfunction in OSA is largely unknown. Endothelial dysfunction in OSA is reversible with antioxidants, suggesting a role for oxidant overproduction in the decreased NO availability in OSA. This provides parallels to other cardiovascular diseases in which oxidative stress induced endothelial dysfunction is important.

Recent studies reported evidence of dysfunction or decreased expression of endothelial nitric oxide synthase (eNOS) in association with increased peroxynitrite in harvested venous endothelial cells of OSA patients. We endeavored to perform the first direct quantification of microvascular endothelial genes from OSA patients. We hypothesized that patients with OSA who are free of any cardiovascular disease will have early functional changes in the microcirculatory endothelial cells that are associated with OSA, and therefore would resolve with treatment. Given the role of oxidative stress in the vascular disease of OSA, we expected to find evidence of superoxide overproduction in the microcirculatory vessels. We expected these functional changes to be reversible with treatment of OSA.

Measurement of superoxide will be done on the subcutaneous biopsy tissue using quantitative Polymerase Chain Reaction (qPCR) and immunohistochemistry techniques and image analysis software. Measurement of endothelial function will be done using Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Completed sleep study - Older than 18

Exclusion Criteria:

* Hypertension
* Diabetes
* coronary disease
* Peripheral vascular disease
* High cholesterol
* Smoking
* Pregnancy
* Use of erectile dysfunction medications or supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People screened for sleep apnea with a completed sleep study who do not have hypertension or coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Khayat, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Patt BT, Jarjoura D, Haddad DN, Sen CK, Roy S, Flavahan NA, Khayat RN. Endothelial dysfunction in the microcirculation of patients with obstructive sleep apnea. Am J Respir Crit Care Med. 2010 Dec 15;182(12):1540-5. doi: 10.1164/rccm.201002-0162OC. Epub 2010 Jul 23. PMID 20656942

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No diagnosis of Obstructive Sleep Apnea or treatment with continuous positive airwary therapy
- Obstructive Sleep Apnea: Participants wear continuous positive airway therapy
Period: Overall Study
Arm/Group | Control | Obstructive Sleep Apnea
Started | 9 | 16
Completed | 9 | 12
Not Completed | 0 | 4
Not completed — failure in cpap compliance | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Obstructive Sleep Apnea | Total
Number analyzed (Participants) | 9 | 16 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 16 | 25
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (7.4) | 43.6 (11.2) | 39.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 12 | 16
Region of Enrollment [Number; unit: participants]
  United States | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation
Description: A non-invasive test using an ultrasound to measure baseline resting vessel diameter and vessel wall dilation in upper arm post application of an inflated blood pressure cuff for five minutes. The percentage change in vessel wall dilation due to stimulation from the resting vessel diameter will be calculated for each group of participants. The results will be compared relative to each group of participants.
Time Frame: Baseline and 12 weeks
Population: Comparative values analyzed for those with endothelial nitric oxide synthase and nitrotyrosine stain density values only.
Measure: Mean (Standard Error); unit: percentage change of vessel diamter
Groups:
- Obstructive Sleep Apnea-pre Treatment: Participants with Obstructive Sleep Apnea prior to receiving positive airway pressure treatment
- Control: Participants with no diagnosis of obstructive sleep apnea and no treatment with continuous positive airway pressure
- Obstructive Sleep Apnea Post Treatment: Participants with Obstructive Sleep Apnea after receiving positive airway pressure treatment for twelve weeks(% dilation change from baseline)
Arm/Group | Obstructive Sleep Apnea-pre Treatment | Control | Obstructive Sleep Apnea Post Treatment
Number analyzed (Participants) | 7 | 7 | 7
percentage change of vessel diamter | 5.7 (.5) | 9.5 (.6) | 7.3 (.9)
Statistical Analysis 1: Comparison: Obstructive Sleep Apnea-pre Treatment vs Obstructive Sleep Apnea Post Treatment; Flow mediated dilation = [(average maximum dilation post cuff deflation - average baseline diameter)/ average baseline diameter]100; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — For comparing pre versus post, paired t tests were used. We considered tests in the hypothesized direction conclusive; For each comparison, we tested at the 0.05 level with double-sided P values. We used no correction for multiple testing when declaring significance

2. Other Pre Specified Outcome: Peroxynitrite Deposition in the Vascular Walls
Description: A forearm biopsy will be collected to isolate human microcirculatory endothelial cells. The stain density of peroxynitrite, an indicator of oxidative stress, in the vascular walls is compared between pre-treatment and post treatment patient tissue. Also another comparison is made between pre-treatment and control tissue. The stain density is a software-generated measurement of pixel intensity and is considered to be an arbitrary unit. Higher numbers indicate greater density
Time Frame: baseline and 12 weeks
Population: Comparative values analyzed for those with endothelial nitric oxide synthase and flow mediated dilation only.
Measure: Mean (Standard Error); unit: stain density units
Groups:
- Obstructive Sleep Apnea-pre Treatment: Participants with Obstructive Sleep Apnea prior to receiving positive airway pressure treatment(Stain Density Units)
- Control: Participants with no diagnosis of obstructive sleep apnea and no treatment with continuous positive airway pressure(Stain Density Units)
- Obstructive Sleep Apnea Post Treatment: Participants with Obstructive Sleep Apnea after receiving positive airway pressure treatment for twelve weeks(Stain Density Units)
Arm/Group | Obstructive Sleep Apnea-pre Treatment | Control | Obstructive Sleep Apnea Post Treatment
Number analyzed (Participants) | 7 | 7 | 7
stain density units | 44.0 (1.6) | 21.8 (1.9) | 30.5 (1.6)
Statistical Analysis 1: Comparison: Obstructive Sleep Apnea-pre Treatment vs Obstructive Sleep Apnea Post Treatment; For comparing pre- versus post-treatment, paired t tests were used. For each variable and comparison, we tested at the 0.05 level with double-sided P values; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — We only consider tests in the hypothesized direction conclusive, so testing is conservative from that perspective. However, we used no correction for multiple testing when declaring significance

ADVERSE EVENTS:
Arm/Group | Control | Obstructive Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/16
Other Adverse Events (participants affected / at risk) | 0/9 | 0/16

LIMITATIONS AND CAVEATS:
Small Feasibility trial only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No